CLINICAL TRIAL: NCT04681612
Title: The Prognostic Role of Indices of Sympathetic Nervous System Overdrive in Patients With Myocardial Infarction With Non-obstructive Coronary Arteries
Brief Title: The Prognostic Role of Indices of Sympathetic Nervous System Overdrive in MINOCA
Acronym: PRISMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hippocration General Hospital (Other)
Collaborators: 401 General Military Hospital of Athens (Other); 251 Hellenic Air Force & VA General Hospital (Other); Athens Naval Hospital (Unknown); Evangelismos General Hospital (Unknown); Aleksandra General Hospital (Unknown); Sismanoglio General Hospital (Other); G.Gennimatas General Hospital (Other); Tzaneio General Hospital of Pireus (Unknown); Elpis General Hospital (Unknown); Thriasio General Hospital of Elefsina (Other); Laiko General Hospital (Unknown); Attikon Hospital (Other); KAT General Hospital (Other)
Responsible Party: Principal Investigator, Konstantinos Tsioufis, Konstantinos Tsioufis, Prof. of Cardiology, Hippocration General Hospital
Other Study IDs: PRISMA-GR
Record Dates: First submitted 2020-12-13; First posted 2020-12-23 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Myocardial Infarction With Nonobstructive Coronary Arteries
Keywords: Myocardial infarction; MINOCA; Sympathetic overdrive; SNS; MSNA; Muscle Microneurography; CMR; Heart rate variability
MeSH Terms: conditions — MINOCA; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples Without DNA — Serum biomarkers Plasma biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MINOCA: Patients hospitalised with MINOCA according to the recently published consensus document of ESC after cardiac MRI confirmation.
  Interventions: Diagnostic Test: MSNA; Diagnostic Test: Heart Rate Variability; Diagnostic Test: Blood Pressure Variability; Diagnostic Test: CMR; Diagnostic Test: History, Lab, clinical and hemodynamic parameters

INTERVENTIONS:
Diagnostic Test: MSNA — Assessed via Muscle Microneurography during the first 14 days of the acute phase.
  Indices: busts/min, busts/100bpm
Diagnostic Test: Heart Rate Variability — Assessed via 24hr ECG monitoring during the first 14 days of the acute phase. Indices: Time-domain, Frequency-domain, Non-linear
Diagnostic Test: Blood Pressure Variability — Assessed via Ambulatory BPM during the first 14 days of the acute phase. Indices: SD, wSD, ARV, CV
Diagnostic Test: CMR — Cardiac Magnetic Resonance during the first 14 days of the acute phase. Assessment of oedema, Late Gadolinium Enhancement ischaemic pattern. Assessment of cardiac function parameters
Diagnostic Test: History, Lab, clinical and hemodynamic parameters — 1. Description of event, 2. Risk factors, 3. Medical history, 4. ECG parameters, 5. ECHO parameters, 6. Hemodynamic parameters of acute phase and hospitalization, 7. Coronary angiogram paraemeters, 7. Complete lab parameter assessment, 8. Thrombofilia assessment, 9. SF-12 QoL and Anxiety and Depression Scale (HADS) questionnaires

SUMMARY:
Myocardial infarction with non-obstructive coronary arteries (MINOCA) occurs in 1-13% of all patients with acute myocardial infarction (AMI). According to most studies MINOCA patients seem to have a more favorable prognosis compared to the obstructive AMI ones, but face a significant risk for recurrent events of angina. It has been demonstrated that sympathetic nervous system (SNS) overdrive during the acute phase of an acute coronary syndrome (ACS) has a deleterious impact on cardiovascular morbidity and mortality and this is the reason why contemporary treatment strategy of ACS aims towards the inhibition of SNS mechanisms. In the setting of MINOCA, however, data are scarce regarding the prognostic role of SNS activation and the concomitant utility of a similar therapeutical approach.

The aim of this study is to investigate the potential role of SNS in cardiovascular prognosis of MINOCA patients. In the same context, this study is the first, to the investigators' knowledge, registry where the working diagnosis of MINOCA will be confirmed with cardiac magnetic resonance (CMR) imaging.

This is an observational cohort study with a prospective follow-up of 18 months enrolling all patients aged 38-85 years old who fulfill the diagnostic criteria of MINOCA. Patients will receive treatment according to the latest guidelines and consensus documents. Assessment of SNS will include calculation of indices of heart rate and blood pressure variability, as well as the measurement of muscle sympathetic nerve activity (MSNA) during the first 14 days following the event. Follow-up will include a phone contact at 3, 6 and 12 months to record potential primary endpoints and a clinic visit at 18 months to reassess clinical and lab parameters and record primary and secondary endpoints. Definition of primary endpoints includes hospitalization for new onset of ACS, heart failure, stroke or transient ischemic attack, cardiovascular death or death from any cause. Secondary endpoints include the burden of arrythmias estimated from 24hr ECG recording, recurrent angina assessed via Seattle Angina Questionnaire (SAQ) and the general health condition and quality of life (QoL) assessed using SF-12 questionnaire.

The results of this study are expected to reveal the prognostic role of SNS assessment in patients with MINOCA with a potential clinical implication in a treatment approach towards the inhibition of SNS mechanisms.

DETAILED DESCRIPTION:
BACKGROUND

Myocardial infarction with non-obstructive coronary arteries (MINOCA) occurs in 1-13% of all patients with acute myocardial infarction (AMI). According to most studies MINOCA patients seem to have a more favorable prognosis compared to the obstructive AMI ones, but face a significant risk for recurrent events of angina. MINOCA consists a clinical entity characterized by a heterogeneous and poorly understood pathophysiological substrate (plaque disruption, coronary epicardial and microvascular spasm, thromboembolism, thrombophilia, spontaneous dissection, myocardial bridges, microvascular dysfunction), whereas current data leave significant knowledge gaps regarding the risk stratification and the proper therapeutical approach of these patients. Sympathetic nervous system (SNS) overdrive during the acute phase of an acute coronary syndrome (ACS) is an expected reflex mechanism aiming to maintain homeostasis. On the other hand, it has been demonstrated that it has a deleterious impact on cardiovascular morbidity and mortality and this is the reason why contemporary treatment strategy of ACS aims towards the inhibition of SNS mechanisms. In the setting of MINOCA, however, data are scarce regarding the prognostic role of SNS activation and the concomitant utility of a similar therapeutical approach.

AIM OF THE STUDY

The primary aim of this study is to investigate the potential role of SNS in cardiovascular prognosis of MINOCA patients. Furthermore, investigators will assess relations between various SNS parameters and clinical characteristics of these patients, as well as other indices of cardiovascular function (biomarkers, imaging). In the same context, this study is the first, to the investigators' knowledge, registry where the working diagnosis of MINOCA will be confirmed with cardiac magnetic resonance (CMR) imaging.

METHODS

This is an observational cohort study with a prospective follow-up of 18 months enrolling all patients aged 35-85 years old who fulfill the diagnostic criteria of MINOCA, on the condition that CMR does not reveal findings compatible with a diagnosis of myocarditis or Takotsubo. Patients will receive treatment according to the latest guidelines and consensus documents. During hospitalization, a complete medical history will be recorded and all basic clinical and lab parameters will be collected. Assessment of SNS will include calculation of indices of heart rate and blood pressure variability derived from 24hr monitoring using validated devices, as well as the measurement of muscle sympathetic nerve activity (MSNA) during the first 14 days following the event. Follow-up will include a phone contact at 3, 6 and 12 months to record potential primary endpoints and a clinic visit at 18 months to reassess clinical and lab parameters and record primary and secondary endpoints. Definition of primary endpoints includes hospitalization for new onset of ACS, heart failure, stroke or transient ischemic attack, cardiovascular death or death from any cause. Secondary endpoints include the burden of arrythmias estimated from 24hr ECG recording, recurrent angina assessed via Seattle Angina Questionnaire (SAQ) and the general health condition and quality of life (QoL) assessed using SF-12 questionnaire and Hospital Anxiety and Depression Scale (HADS).

- Sympathetic tone estimation:

Α. MSNA. After patient's stabilization the test will be performed and the derived data will be the number of bursts per min and the average bursts per 100 beats.

B. Ambulatory heart rate and blood pressure monitoring. Heart rate variability will be analyzed via Kubios software for short-term and long-term heart rate variability. Blood pressure short-term variability will be expressed as SD, wSD, ARV, CV, time rate of BP variation.

For data analysis, SPSS 24.0 software will be used. Continuous parametric data will be expressed as mean and SD. For categoric parametric data results will be presented in means of frequency and percentage. Comparisons between categoric parameters will be done with test x2. Comparisons between the mean values for continuous parameters with normal distribution will be done via unpaired student's test. Comparisons between categoric parameters will be done with Mann Whitney U test. Normal distribution will be checked with Kolmogorov-Smirnov test. Correlation analysis will be done via Pearson Phi coefficient or Spearman Rho. Statistically significant will be differences with p value < 0.05. Evaluation of correlations between selected variables and cardiovascular events and mortality will be via Kaplan Maier curves.

STUDY LIMITATIONS

* Study will include MINOCA patients irrespective of the underlying pathophysiological mechanism. This is the result of the inablity of most centers to perform intravascular imaging (IVUS, OCT) on a routine basis and the tendency to avoid spasm provoking procedures during coronary angiography.
* Although most data will be recorded during the acute/hospitalization phase, the time frame of MSNA and CMR is expected to vary according to the clinical state of the participants and the technical capabilities of the centers. However, an effort will be made not to overlap the 14 days time limit proposed by the majority of investigators.
* CMR will be take place in different centers thus some extent of interobserver variability is expected. However results will be reassessed by a single investigator.

ESTIMATED RESEARCH OUTCOMES

* It will be the first registry, to the investigators' knowledge, that will record data of SNS activation in patients will CMR-confirmed MINOCA.
* The results of the present study are expected to reveal the prognostic role of SNS assessment in patients with MINOCA with a potential clinical implication in a treatment approach towards the inhibition of SNS mechanisms.
* Furthermore, assessment of correlations between parameters of cardiac function and CMR imaging with the level of SNS activation will provide a valuable insight towards the elucidation of the potential role of SNS overdrive during the acute phase of MINOCA.
* Last but not least, follow up assessment will provide information regarding the long-term incidence of persistent or recurrent angina as well as the impact of MINOCA in future quality of life, sentimental state and general health status.

ELIGIBILITY:
Inclusion Criteria:

* Patients 35-85 years old.
* Signed ICF.
* Cases fulfilling the MINOCA criteria according to working group position paper and after CMR confirmation of ischemic pattern LGE (excluding myocarditis and Takotsubo)

Exclusion Criteria:

* Age <35 and >85 years old
* Myocarditis or Takotsubo (CMR confirmation)
* No CMR available (CKD stage IV-V, pacemaker)
* Inability to assess SNS (polyneuropathy, peripheral neuropathy, dysautonomy, permanent AF)
* Severe valvular disease
* LVEF<35%
* Life expenctancy less than the follow up period on recruitement
* Active cancer on treatment
* Psychiatric illness compromising follow up

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with MINOCA according to working group position paper and after CMR confirmation of ischemic pattern LGE (excluding myocarditis and Takotsubo)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence (%) of Death during follow up | Assessed at 4 time points after the acute event: 3 months, 6 months, 12 months, 18 months
  Number of participants dead due to cardiovascular or any other cause
Incidence (%) of Hospitalization for Major Cardiovascular Events (MACEs) during follow up | Assessed at 4 time points after the acute event: 3 months, 6 months, 12 months, 18 months
  Number of participants hospitalized due to: ACS (STEMI,NSTEMI,Unstable Angina), Decompensated heart failure, Stroke
Incidence (%) of the Composite endpoint | Assessed at 4 time points after the acute event: 3 months, 6 months, 12 months, 18 months
  Incidence (%) of the composite endpoint that includes: Number of participants either hospitalized for MaCEs (ACS, Decompensated heart failure, Stroke) or dead due to a cardiovascular or any other cause

SECONDARY OUTCOMES:
Frequency (%) of increased long term arrythmia burden | Assessed at 18 months after the acute event
  Number of participants fulfilling 1 or more criteria for increased arrythmia burden assessed via 24hr ECG monitor at follow up visit.
  Criteria assessed: PVCs>10%, AF>30sec, NSVT, complete heart block
Frequency of long term Sustained/ Reccurent Angina | Assessed at 18 months after the acute event
  Seattle angina questionnaire (SAQ) will be filled by participants at follow up visit.
  SAQ provides a quantification of sentimental and physical impact of angina on participants. It is a 19-question self-administered questionnaire assessing physical limitation, angina persistence and frequency, satisfaction of treatment and the overall impact of the disease on the participant. Scores range from 0 to 100. Lower scores depict a greater overall impact of angina on the participant.
Assessment of Quality of Life and General Health Status | Assessed at 1-14 days and 18 months after the acute event
  Medical Outcomes Study 12-Item Short Form (SF-12) will be filled by participants during the acute phase and follow up visit in order to assess the long term impact of MINOCA on the participants' quality of life. SF-12 consists of 12 questions and its score ranges from 0 to 100. Lower scores depict a worse quality of life for the participant.
Assessment of Sentimental status | Assessed at 1-14 days and 18 months after the acute event
  Hospital Anxiety and Depresion Scale (HADS) questionnaire will be filled by participants during the acute phase and follow up visit in order to assess the long term impact of MINOCA on the participants' emotional status (anxiety, depression). HADS consists of 14 questions and its score ranges from 0 to 21 separetely for anxiety and depression quantification.
  Scores: 0-7 = Normal, 8-10 = Borderline abnormal (borderline case), 11-21 = Abnormal (case).

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil K. Mantzouranis, MD, Study Director — Hippokration Hospital; Ioannis E. Leontsinis, MD, Study Director — Hippokration Hospital
Locations (1):
- Hippokration Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pasupathy S, Tavella R, Beltrame JF. The What, When, Who, Why, How and Where of Myocardial Infarction With Non-Obstructive Coronary Arteries (MINOCA). Circ J. 2016;80(1):11-6. doi: 10.1253/circj.CJ-15-1096. Epub 2015 Nov 20. PMID 26597354
- [Background] Tamis-Holland JE, Jneid H, Reynolds HR, Agewall S, Brilakis ES, Brown TM, Lerman A, Cushman M, Kumbhani DJ, Arslanian-Engoren C, Bolger AF, Beltrame JF; American Heart Association Interventional Cardiovascular Care Committee of the Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; and Council on Quality of Care and Outcomes Research. Contemporary Diagnosis and Management of Patients With Myocardial Infarction in the Absence of Obstructive Coronary Artery Disease: A Scientific Statement From the American Heart Association. Circulation. 2019 Apr 30;139(18):e891-e908. doi: 10.1161/CIR.0000000000000670. PMID 30913893
- [Background] Agewall S, Beltrame JF, Reynolds HR, Niessner A, Rosano G, Caforio AL, De Caterina R, Zimarino M, Roffi M, Kjeldsen K, Atar D, Kaski JC, Sechtem U, Tornvall P; WG on Cardiovascular Pharmacotherapy. ESC working group position paper on myocardial infarction with non-obstructive coronary arteries. Eur Heart J. 2017 Jan 14;38(3):143-153. doi: 10.1093/eurheartj/ehw149. No abstract available. PMID 28158518
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Background] Pasupathy S, Air T, Dreyer RP, Tavella R, Beltrame JF. Systematic review of patients presenting with suspected myocardial infarction and nonobstructive coronary arteries. Circulation. 2015 Mar 10;131(10):861-70. doi: 10.1161/CIRCULATIONAHA.114.011201. Epub 2015 Jan 13. PMID 25587100
- [Background] Lindahl B, Baron T, Erlinge D, Hadziosmanovic N, Nordenskjold A, Gard A, Jernberg T. Medical Therapy for Secondary Prevention and Long-Term Outcome in Patients With Myocardial Infarction With Nonobstructive Coronary Artery Disease. Circulation. 2017 Apr 18;135(16):1481-1489. doi: 10.1161/CIRCULATIONAHA.116.026336. Epub 2017 Feb 8. PMID 28179398
- [Background] Dreyer RP, Tavella R, Curtis JP, Wang Y, Pauspathy S, Messenger J, Rumsfeld JS, Maddox TM, Krumholz HM, Spertus JA, Beltrame JF. Myocardial infarction with non-obstructive coronary arteries as compared with myocardial infarction and obstructive coronary disease: outcomes in a Medicare population. Eur Heart J. 2020 Feb 14;41(7):870-878. doi: 10.1093/eurheartj/ehz403. PMID 31222249
- [Background] Grodzinsky A, Arnold SV, Gosch K, Spertus JA, Foody JM, Beltrame J, Maddox TM, Parashar S, Kosiborod M. Angina Frequency After Acute Myocardial Infarction In Patients Without Obstructive Coronary Artery Disease. Eur Heart J Qual Care Clin Outcomes. 2015;1(2):92-99. doi: 10.1093/ehjqcco/qcv014. Epub 2015 Jul 23. PMID 28239487
- [Background] Tsioufis C, Iliakis P, Kasiakogias A, Konstantinidis D, Lovic D, Petras D, Doumas M, Tsiamis E, Papademetriou V, Tousoulis D. Non-pharmacological Modulation of the Autonomic Nervous System for Heart Failure Treatment: Where do We Stand? Curr Vasc Pharmacol. 2017;16(1):30-43. doi: 10.2174/1570161115666170428124756. PMID 28462724
- [Background] Jamali HK, Waqar F, Gerson MC. Cardiac autonomic innervation. J Nucl Cardiol. 2017 Oct;24(5):1558-1570. doi: 10.1007/s12350-016-0725-7. Epub 2016 Nov 14. PMID 27844333
- [Background] Parati G, Ochoa JE, Lombardi C, Bilo G. Assessment and management of blood-pressure variability. Nat Rev Cardiol. 2013 Mar;10(3):143-55. doi: 10.1038/nrcardio.2013.1. Epub 2013 Feb 12. PMID 23399972
- [Background] Stergiou GS, Kollias A, Ntineri A. Assessment of drug effects on blood pressure variability: which method and which index? J Hypertens. 2014 Jun;32(6):1197-200. doi: 10.1097/HJH.0000000000000201. No abstract available. PMID 24781510
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Arsenos P, Gatzoulis K, Dilaveris P, Manis G, Tsiachris D, Archontakis S, Vouliotis AI, Sideris S, Stefanadis C. Arrhythmic sudden cardiac death: substrate, mechanisms and current risk stratification strategies for the post-myocardial infarction patient. Hellenic J Cardiol. 2013 Jul-Aug;54(4):301-15. No abstract available. PMID 23912922
- [Background] Liao D, Carnethon M, Evans GW, Cascio WE, Heiss G. Lower heart rate variability is associated with the development of coronary heart disease in individuals with diabetes: the atherosclerosis risk in communities (ARIC) study. Diabetes. 2002 Dec;51(12):3524-31. doi: 10.2337/diabetes.51.12.3524. PMID 12453910
- [Background] Vallbo AB, Hagbarth KE, Wallin BG. Microneurography: how the technique developed and its role in the investigation of the sympathetic nervous system. J Appl Physiol (1985). 2004 Apr;96(4):1262-9. doi: 10.1152/japplphysiol.00470.2003. PMID 15016790
- [Background] Shoemaker JK, Klassen SA, Badrov MB, Fadel PJ. Fifty years of microneurography: learning the language of the peripheral sympathetic nervous system in humans. J Neurophysiol. 2018 May 1;119(5):1731-1744. doi: 10.1152/jn.00841.2017. Epub 2018 Feb 7. PMID 29412776